CLINICAL TRIAL: NCT02403206
Title: Femtosecond Laser Assisted Cataract Surgery in Intumescent Cataracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTW860-P001
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-06

CONDITIONS: Intumescent Cataract
MeSH Terms: interventions — Capsulorhexis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Laser (Experimental): Femtosecond laser assisted capsulotomy and corneal incision performed during cataract surgery
  Interventions: Device: Femtosecond laser
- Manual (Active Comparator): Continuous curvilinear capsulorhexis performed during cataract surgery
  Interventions: Procedure: Continuous Curvilinear Capsulorhexis (CCC)

INTERVENTIONS:
Device: Femtosecond laser — Laser console and a patient interface used to cut tissue during cataract removal of the crystalline lens
  Other Names: LenSx® Laser
  Arms: Laser
Procedure: Continuous Curvilinear Capsulorhexis (CCC) — Standard-of care manual procedure (using either needles or forceps) for creating capsulorhexis, ie., opening in capsular bag during anterior segment ophthalmic surgery
  Arms: Manual

SUMMARY:
The purpose of the study is to compare femtosecond laser-assisted capsulotomy to manual capsulorhexis in patients with intumescent cataracts. An intumescent cataract is defined as a cataract with a pressurized capsular bag.

ELIGIBILITY:
Inclusion Criteria:

* Willing to undergo cataract surgery.
* Able to lie flat in a supine position.
* Able to understand and willing to sign the Informed Consent Form (ICF).
* Presenting with intumescent white cataract, with a liquid pressurized bag and a milky, liquid cortex.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Pregnant or lactating mothers.
* Corneal disease that precludes application of the cornea or transmission of laser light at 1030 nanometer (nm) wavelength.
* Corneal opacity that would interfere with the laser beam.
* Presence of blood or other material in the anterior chamber.
* Hypotony or presence of corneal implant.
* Poorly dilating pupils.
* Condition which would cause inadequate clearance between the intended capsulotomy depth and the endothelium.
* Residual, recurrent, active ocular or eye lid disease, including any corneal abnormality.
* Any contraindication to cataract surgery.
* Other protocol-specified exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Surgical, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 14 investigative sites: 1 located in Greece, 4 located in India, 2 located in Mexico, 1 located in the Philippines, 3 located in Romania, and 3 located in the US.
Pre-assignment Details: Of the 406 enrolled, 6 subjects were exited as screen failures and 10 withdrew prior to randomization. This reporting group includes all randomized subjects (390).
Groups:
- Laser (LSX): Femtosecond laser assisted capsulotomy and corneal incision performed during cataract surgery
- Manual (CCC): Continuous curvilinear capsulorhexis (CCC) performed during cataract surgery
Period: Overall Study
Arm/Group | Laser (LSX) | Manual (CCC)
Started | 194 | 196
Treated Prior to Randomization | 0 | 1
Randomized and Treated | 188 | 190
Completed | 183 | 186
Not Completed | 11 | 10
Not completed — Lost to Follow-up | 4 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Reason not given | 2 | 4

BASELINE CHARACTERISTICS:
Population: This analysis population includes subjects who signed an informed consent form, were randomized, and underwent the removal of an intumescent cataract with subsequent IOL implantation (Intent-to-Treat (ITT)).
Groups:
- Manual (CCC): CCC performed during cataract surgery
- Total: Total of all reporting groups
Arm/Group | Laser (LSX) | Manual (CCC) | Total
Number analyzed (Participants) | 187 | 189 | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (13.6) | 66.4 (11.9) | 65.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 117 | 227
  Male | 77 | 72 | 149

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Capsular Tears (Anterior or Posterior) During Surgery
Description: A capsular tear is defined as any unintended tear on the anterior or posterior capsule and includes a radial tear that moves peripherally on the anterior capsule during capsulotomy and extends to form a posterior capsular tear during intumescent cataract surgery. An intumescent cataract is defined as a cataract with a pressurized capsular bag. A lower value indicates fewer capsular tears. Only one eye (study eye) contributed to the analysis.
Time Frame: Day 0 (operative day)
Population: Intent-to-Treat Analysis Set
Measure: Number; unit: percentage of capsular tears
Arm/Group | Laser (LSX) | Manual (CCC)
Number analyzed (Participants) | 187 | 189
percentage of capsular tears | 5.3 | 5.3

2. Secondary Outcome: Operating Time in the Eye to Complete Entire Cataract Procedure
Description: Operating time in the eye was the time interval (in seconds) from the time the corneal incision was opened to the time the wound was closed. Only one eye (study eye) contributed to the analysis.
Time Frame: Day 0 (operative day)
Population: Intent-to-Treat Analysis Set
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Laser (LSX) | Manual (CCC)
Number analyzed (Participants) | 187 | 189
seconds | 795.0 (354.7) | 856.6 (436.3)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 75 days). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational product (test or control article). AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- Pretreatment: All subjects who consented to participate in the study prior to initiation of study treatment
- Laser (LSX): Subjects who underwent femtosecond laser-assisted cataract surgery
- Manual (CCC): Subjects who underwent CCC-assisted cataract surgery
Arm/Group | Pretreatment | Laser (LSX) | Manual (CCC)
All-Cause Mortality (participants affected / at risk) | 0/406 | 0/188 | 0/191
Serious Adverse Events (participants affected / at risk) | 1/406 | 16/188 | 14/191
Other Adverse Events (participants affected / at risk) | 0/406 | 46/188 | 43/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=406) | Laser (LSX) (N=188) | Manual (CCC) (N=191)
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Aphakia (Eye disorders) | 0 | 0 | 1
Iridocele (Eye disorders) | 0 | 0 | 1
Iris adhesions (Eye disorders) | 0 | 0 | 1
Iris atrophy (Eye disorders) | 0 | 0 | 1
Posterior capsule rupture (Eye disorders) | 0 | 4 | 2
Retinal detachment (Eye disorders) | 0 | 0 | 1
Vitreous loss (Eye disorders) | 0 | 2 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 9 | 9
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Eye operation (Surgical and medical procedures) | 0 | 2 | 0
Glaucoma surgery (Surgical and medical procedures) | 0 | 1 | 0
Intraocular lens implant (Surgical and medical procedures) | 0 | 0 | 1
Retinopexy (Surgical and medical procedures) | 0 | 0 | 1
Vitrectomy (Surgical and medical procedures) | 1 | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=406) | Laser (LSX) (N=188) | Manual (CCC) (N=191)
Conjunctival haemorrhage (Eye disorders) | 0 | 11 | 2
Corneal disorder (Eye disorders) | 0 | 16 | 19
Corneal oedema (Eye disorders) | 0 | 40 | 39
Ocular hypertension (Eye disorders) | 0 | 10 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.